CLINICAL TRIAL: NCT03896867
Title: Anapod™ Humi-Therm Heated Humidification System Breathing Circuit Versus Bair Hugger™ Warming Blanket for Intraoperative Maintenance of Body Temperature in Pediatric Patients Undergoing Dental Procedures: a Prospective Randomized Non-Inferiority Study
Brief Title: Heated Humidification System Breathing Circuit for Maintenance of Body Temperature in Pediatric Patients
Acronym: ANAPOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ANES-2019-27433
Record Dates: First submitted 2019-03-21; First posted 2019-04-01 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Temperature Change, Body
Keywords: Temperature management; Perioperative temperature management; Pediatric temperature management; Pediatric perioperative temperature management
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Group assignment will be blinded with the data set (Group A vs B) for review purposes - although it is important to note that true blinding of the providers (including on PI and Co PI) is impossible for this procedural study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Anapod™ Humi-Therm Heated Humidification System (Experimental): Patient warming will be provided via the Anapod™ Humi-Therm Heated Humidification System Breathing Circuit.
  Interventions: Device: Anapod™ Humi-Therm Heated Humidification System Breathing Circuit
- Bair Hugger™ Warming Blanket (Active Comparator): Patient warming will be provided via the Bair Hugger™ Warming Blanket.
  Interventions: Device: Bair Hugger™ Warming Blanket

INTERVENTIONS:
Device: Anapod™ Humi-Therm Heated Humidification System Breathing Circuit — For the Anapod™ group, the BairHugger™ blanket will be connected, but the unit will not be turned on. The Anapod™ will be used with a starting circuit temperature set at the standard 45°C (note, this is temperature at the unit - NOT the temperature of the gas reaching the trachea). In the event that the patient's rectal temperature falls below 35.6C, the BairHugger™ warming system will be activated ("Hypothermic Rescue"). In the event that rectal temperature increases to a value of ≥37.5C, the Anapod system will be turned off - and the BairHugger turned on with the warming unit set to "ambient" (meaning cool operating room temperature will be blown over the patient ("Hyperthermic Rescue").
  Arms: Anapod™ Humi-Therm Heated Humidification System
Device: Bair Hugger™ Warming Blanket — For the BairHugger™ group, the blanket will be used with a starting temperature set at HIGH. The BairHugger™ unit will be attached to the warming unit and started as soon as possible. In the event that the patient's rectal temperature falls below 35.6C, the Anapod™ warming system will be activated ("Rescue"). In the event that rectal temperature increases to a value of ≥37.5C, the BairHugger™ warming unit will be set to "ambient" (meaning cool operating room temperature will be blown over the patient ("Hyperthermic Rescue").
  Arms: Bair Hugger™ Warming Blanket

SUMMARY:
Our goal is to evaluate the efficacy of the Westmed system vs the Bair Hugger Blanket.

DETAILED DESCRIPTION:
Temperature management is an important aspect of perioperative care that falls under the purview of the anesthesiologist. Temperature is recognized as one of four primary vital signs and significant deviations from normal values may result in patient harm. General anesthesia disrupts the body's temperature homeostasis by inhibiting temperature regulation mechanisms such as vasoconstriction/-dilation, shivering and behavioral interventions (donning clothes or leaving an area with excessive heat, for example). Anesthetized patient have a tendency to become hypothermic, especially during long surgical procedures. This results from both the redistribution of cooler peripheral temperatures into the core (due to vasodilation) as well as actual temperature loss to a cold operating room environment (which is maintained at a lower temperature for the comfort of fully gowned surgeons and nurses). In addition, large surgical incisions predispose the patient to hypothermia through evaporation and convection.

Hypothermia is a recognized risk factor that predisposes the patient to an increased metabolic rate, increased oxygen demand, coagulopathies, impaired wound healing, impaired immune function and increased risk of infection. Therefore, maintenance of normal body temperature is an important goal of every general anesthetic - and is a well-accepted quality metric associated with patient care. Because of the greater surface area to volume relationship, children are thought to be a greater risk of intraoperative hypothermia.

The most widely used method of maintaining body temperature during surgery (and a routine at this institution) is by using a forced-air warming blanket (Bair Hugger warming blanket, 3M). Despite its widespread use, the forced-air warming blanket has its limitations. For example, during certain surgical procedures, the location of the surgical field precludes placement of the warming blanket. In addition, the warming blanket often cannot be placed immediately after the induction of anesthesia (when complex patient positioning is required) - leaving the patient exposed to hypothermic conditions for short (10-15min) or long (30-60min) periods of time. There is hence a need for alternative warming systems that could be implemented immediately following anesthetic induction.

Westmed, Inc. has developed an alternative system that utilizes a heated, humidified breathing circuit to regulate a patient's body temperature in the intraoperative setting. This system is active from the moment the trachea is intubated following anesthetic induction, i.e. there are no delays in instituting thermal management.

ELIGIBILITY:
Inclusion Criteria:

- Pediatric patients undergoing elective, scheduled dental procedures at Masonic Children's hospital requiring general anesthesia with endotracheal intubation, anticipated to last 1-6 hours or longer

Exclusion Criteria:

* Parent refusal of consent
* Patient refusal of assent (if applicable)
* Additional procedures (combined procedures) that involve other specialties besides dentists and other parts of the patient's body other than the oral cavity.
* History of diseases associated with temperature dysregulation (active hyperthyroidism, dysautonomia, osteogenesis imperfecta, history of malignant hyperthermia)
* Patients that will not be intubated for the procedure

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anapod™ Humi-Therm Heated Humidification System | Bair Hugger™ Warming Blanket
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anapod™ Humi-Therm Heated Humidification System | Bair Hugger™ Warming Blanket | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 29 | 30 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 6 | 20
  White | 22 | 25 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Rectal Temperature
Description: Last measured core temperature at conclusion of the procedure (measured with rectal temperature probe) in patients assigned to the two warming systems.
Time Frame: study visit 1, at conclusion of dental procedure/anesthesia administration, approximately 1-6 hours
Measure: Mean (Standard Deviation); unit: degrees celsius
Arm/Group | Anapod™ Humi-Therm Heated Humidification System | Bair Hugger™ Warming Blanket
Number analyzed (Participants) | 50 | 50
degrees celsius | 36.7 (0.47) | 37.2 (0.38)

2. Secondary Outcome: Need for Hyperthermic or Hypothermic Rescue
Description: Procedures for hyperthermic and hypothermic rescue can be found in the arm description section. Total number of rescue events will be compared between groups. A greater number of events indicates worse performance for that temperature control method.
Time Frame: study visit 1, measured continuously throughout dental procedure/anesthesia administration, approximately 1-6 hours
Measure: Number; unit: rescue events
Arm/Group | Anapod™ Humi-Therm Heated Humidification System | Bair Hugger™ Warming Blanket
Number analyzed (Participants) | 50 | 50
rescue events | 11 | 22

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | Anapod™ Humi-Therm Heated Humidification System | Bair Hugger™ Warming Blanket
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 12/50 | 25/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anapod™ Humi-Therm Heated Humidification System (N=50) | Bair Hugger™ Warming Blanket (N=50)
prolonged hospitalization (General disorders) | 1 (1) | 2 (2)
Hypothermia (General disorders) | 8 (8) | 1 (1)
Hyperthermia (General disorders) | 3 (3) | 21 (21)
Viral Illness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT03896867/Prot_SAP_001.pdf